CLINICAL TRIAL: NCT02133742
Title: A PHASE 1B, OPEN LABEL, DOSE FINDING STUDY TO EVALUATE SAFETY, PHARMACOKINETICS AND PHARMACODYNAMICS OF AXITINIB (AG-013736) IN COMBINATION WITH PEMBROLIZUMAB (MK-3475) IN PATIENTS WITH ADVANCED RENAL CELL CANCER
Brief Title: A Dose Finding Study To Evaluate Safety, Drug Interaction, Tumor Markers Of Axitinib In Combination With MK-3475 In Adult Patients With Previously Untreated Advanced Renal Cell Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Masking: None | Purpose: Treatment
Other Study IDs: A4061079; KN-035 (Other: Merck)
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Renal Cell Carcinoma
Keywords: Axitinib and MK-3475; patients with advanced Renal Cell Cancer.
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose finding phase and dose expansion phase (Experimental): To test the maximum tolerated dose of MK-3475 at 2 mg/kg every three weeks intravenous infusion in combination with approved axitinib dose
  Interventions: Drug: Axitinib; Drug: MK-3475

INTERVENTIONS:
Drug: Axitinib — Axitinib at starting dose of 5 mg and 3 mg BID.
Drug: MK-3475 — MK-3475 with two dose levels: 2 mg/kg every three weeks to find the maximum tolerated dose and continue treatment in a dose expansion phase.

SUMMARY:
Despite substantial improvements of patients outcome in advanced RCC, durable and complete response is uncommon. The majority of patients eventually develop resistance and exhibit disease progression. Combining a PD-1 inhibitor, which has shown single-agent efficacy with axitinib may provide additional clinical benefit compared to axitinib alone.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced RCC with predominantly clear-cell subtype with primary tumor resected
* At least one measureable lesion as defined by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
* Eastern Cooperative Oncology Group performance status 0 or 1
* Controlled hypertension

Exclusion Criteria:

* Prior treatment with systemic therapy for advanced RCC
* Prior adjuvant or neoadjuvant therapy if disease progression or relapse has occurred during or within 12 months after the last dose of treatment
* Prior treatment with any agent specifically targeting T-cell co-stimulation or checkpoint pathways
* Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis
* Diagnosis of any non-RCC malignancy occurring within 2 years prior to the date of randomization except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or of the cervix or low grade prostate cancer with no plans for treatment intervention
* In past 12 months: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack
* In past 6 months: deep vein thrombosis or pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2019-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (19):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center & Research Institute, Inc., Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Attn. Alicia Sammarco, RPh, NYU Investigational Pharmacy, New York, New York
  - NYU Langone Medical Center, New York, New York
  - NYU Langone, New York, New York
  - Investigational Drug Services, Columbus, Ohio
  - James Cancer Hospital, Columbus, Ohio
  - The Ohio State University Brain and Spine Hospital, Columbus, Ohio
  - Martha Morehouse Medical Plaza, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Vanderbilt Oncology Pharmacy, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Atkins MB, Plimack ER, Puzanov I, Fishman MN, McDermott DF, Cho DC, Vaishampayan U, George S, Tarazi JC, Duggan W, Perini R, Thakur M, Fernandez KC, Choueiri TK. Axitinib plus pembrolizumab in patients with advanced renal-cell carcinoma: Long-term efficacy and safety from a phase Ib trial. Eur J Cancer. 2021 Mar;145:1-10. doi: 10.1016/j.ejca.2020.12.009. Epub 2021 Jan 4. PMID 33412465
- [Derived] Martini JF, Plimack ER, Choueiri TK, McDermott DF, Puzanov I, Fishman MN, Cho DC, Vaishampayan U, Rosbrook B, Fernandez KC, Tarazi JC, George S, Atkins MB. Angiogenic and Immune-Related Biomarkers and Outcomes Following Axitinib/Pembrolizumab Treatment in Patients with Advanced Renal Cell Carcinoma. Clin Cancer Res. 2020 Nov 1;26(21):5598-5608. doi: 10.1158/1078-0432.CCR-20-1408. Epub 2020 Aug 18. PMID 32816890
- [Derived] Atkins MB, Plimack ER, Puzanov I, Fishman MN, McDermott DF, Cho DC, Vaishampayan U, George S, Olencki TE, Tarazi JC, Rosbrook B, Fernandez KC, Lechuga M, Choueiri TK. Axitinib in combination with pembrolizumab in patients with advanced renal cell cancer: a non-randomised, open-label, dose-finding, and dose-expansion phase 1b trial. Lancet Oncol. 2018 Mar;19(3):405-415. doi: 10.1016/S1470-2045(18)30081-0. Epub 2018 Feb 10. PMID 29439857
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061079&StudyName=A%20Phase%201b%2C%20Open%20Label%2C%20Dose%20Finding%20Study%20To%20Evaluate%20Safety%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Axitinib%20%28ag-013736%29%20In%20Combination%20With%20Pembrolizumab%20%28mk-3475%29%20In%20Patients%20With%20Advanced%20Renal%20Cell%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was planned to be conducted in two potential doses in the dose finding phase, Axitinib 3 mg + Pembrolizumab (MK-3475) 2 mg and Axitinib 5 mg + MK 3475 2 mg. However, no participant was enrolled in the Axitinib 3 mg + MK-3475 2 mg reporting group and all participants were enrolled in ''Axitinib 5 mg + MK-3475 2 mg'' reporting group only.
Groups:
- Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg: Participants with no prior systemic treatment for advance cancer, received axitinib 5 mg twice daily orally in combination with pembrolizumab (MK-3475) 2 mg/kg of body weight intravenous infusion every 3 weeks up to a maximum of 6 months in dose finding phase (each cycle of 21 days). Participants received axitinib up to a maximum of 64 cycles and pembrolizumab up to 56 cycles in dose expansion phase (each cycle of 21 days) until documented disease progression or unacceptable toxicity or study discontinuation criteria were met.
Period: Period 1: Dose Finding Phase (6 Months)
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Started | 11
Completed | 11
Not Completed | 0
Period: Period 2:Dose Expansion Phase (1344days)
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Started | 52 (Participants participated in dose finding phase continued treatment in dose expansion phase.)
Completed | 0
Not Completed | 52
Not completed — Lost to Follow-up | 2
Not completed — End of survival follow-up/treatment | 31
Not completed — Death | 13
Not completed — Participant refused further follow-up | 5
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all enrolled participants in dose finding and dose expansion phases who received at least 1 dose of axitinib or pembrolizumab.
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 45
  Black | 1
  Asian | 4
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLT): Dose Finding Phase
Description: DLT was defined as any of the following adverse events (AEs) occurring in the first two cycles of treatment which were attributable to one or both the study drugs: 1) Grade 4 neutropenia, 2) Febrile neutropenia lasting greater than (>) 1 hour, 3) Grade greater than or equal to (>=) 3 neutropenia with infection, 4) Grade >=3 thrombocytopenia with bleeding, 4) Grade 4 thrombocytopenia, 5) Any grade >=3 non-hematologic: non-laboratory toxicities despite maximum supportive therapy or hypertension despite maximal medical therapy, 6) Grade >=3 non-hematologic toxicities resulted in hospitalisation or medical intervention 7) Inability to complete at least 75 percent (%) of axitinib dosing or 2 infusions of pembrolizumab within the DLT observation period (up to 42 days) due to treatment related toxicity. Severity of AEs was graded according to NCI (National Cancer Institute) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: Cycle 1 Day 1 to Cycle 2 Day 21 (up to 42 days)
Population: Per protocol analysis set included all enrolled eligible participants who received at least 1 dose of axitinib or pembrolizumab and experienced DLT during first 2 cycles, or complete the observation period for first 2 cycles of treatment. Here, number of participant analyzed (N) = number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Axitinib 5 mg + Pembrolizumab 2 mg: Dose Finding Phase: Participants with no prior systemic treatment for advance cancer, received axitinib 5 mg twice daily orally in combination with pembrolizumab (MK-3475) 2 mg/kg of body weight intravenous infusion every 3 weeks up to a maximum of 6 months in dose finding phase (each cycle of 21 days).
Arm/Group | Axitinib 5 mg + Pembrolizumab 2 mg: Dose Finding Phase
Number analyzed (Participants) | 11
Participants | 3

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant and jeopardized the participants or required treatment to prevent other AE outcomes for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs are events which occurred between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to 28 days after last dose of study drug (approximately up to 1552 days)
Population: Safety analysis set included all enrolled participants who received at least one dose of axitinib or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
Participants
  AEs | 52
  SAEs | 29

3. Secondary Outcome: Number of Participants With Treatment Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant and jeopardized the participants or required treatment to prevent other AE outcomes for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs are events which occurred between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. Relatedness to study drug was assessed by the investigator.
Time Frame: Baseline up to 28 days after last dose of study drug (approximately up to 1552 days)
Population: Safety analysis set included all enrolled participants who received at least one dose of axitinib or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
Participants
  AEs | 52
  SAEs | 23

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) According to Severity of Grade 3 or Higher Severity Based on NCI CTCAE Version 4.03
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant and jeopardized the participants or required treatment to prevent other AE outcomes for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs were graded according to the Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03 and coded using the Medical Dictionary for Regulatory Activities (MedDRA) as Grade 3: Severe, Grade 4: Life threatening, Grade 5: Death related to AE. Participants were counted once according to the maximum grade observed.
Time Frame: Baseline up to 28 days after last dose of study drug (approximately up to 1552 days)
Population: Safety analysis set included all enrolled participants who received at least one dose of axitinib or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
Participants
  Grade 3 or 4 | 38
  Grade 5 | 1

5. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities of Grade 3 or Higher Severity Based on NCI CTCAE Version 4.03: Biochemistry and Hematology
Description: Laboratory parameters included hematological and biochemistry parameters. Biochemistry parameters included alanine aminotransferase, alkaline phosphatase, aspartate aminotransferase, bilirubin (total), creatinine, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, hypophosphatemia. Hematology parameters included anemia, haemoglobin increased, lymphocyte count increased, lymphopenia, neutrophils (absolute), platelets and white blood cells. Test abnormalities were graded by NCI CTCAE version 4.03 as Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Only categories with at least 1 participant with abnormality are reported in this outcome measure.
Time Frame: Baseline up to a maximum of 1083 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
Participants
  Alanine aminotransferase: Grade 3 | 2
  Hypercalcemia: Grade 3: number analyzed (Participants) | 51
  Hypercalcemia: Grade 3 | 1
  Hyperglycemia: Grade 3 | 5
  Hyperkalemia: Grade 3 | 1
  Hypermagnesemia; Grade 3 | 1
  Hypokalemia: Grade 3 | 3
  Hyponatremia: Grade 3 | 4
  Hypophosphatemia: Grade 3 | 7
  Lymphopenia: Grade 3 | 4
  Neutrophils (absolute): Grade 3 | 2

6. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities: Urinalysis
Description: Urinalysis parameter included urine protein, urine blood/hemoglobin and urine glucose. Test abnormalities was defined as deviation from normal range. Normal range of 24-hour urine protein test: less than 150 mg of protein per day, urine glucose: 0 to 0.8 mmol/L (millimoles per liter), urine protein: 0 to 20 mg/dL (milligrams per deciliter). Urine blood/hemoglobin abnormality was defined as presence and absence of blood/hemoglobin in urine of participants.
Time Frame: Baseline up to a maximum of 1083 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
Participants
  Urine protein (24 hrs) | 0
  Urine blood/hemoglobin | 11
  Urine glucose | 9
  Urine protein | 25

7. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included blood pressure, pulse rate and weight. Change from baseline values were considered to be clinically significant based on investigator's judgement.
Time Frame: Baseline up to a maximum of 1083 days
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
Participants | 0

8. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group [ECOG] Performance Status Score
Description: ECOG performance status was used to assess how disease affect the daily living abilities of a participant. It was measured on a scale ranging from 0 to 4, where 0=fully active (able to carry on all pre-disease activities without restriction); 1=restricted in physically strenuous activity but ambulatory (able to carry out light/sedentary work); 2=ambulatory and capable of all self-care but unable to carry out any work activities (for more than 50% of waking hours); 3=capable of limited self-care, confined to bed or chair (for >50% of waking hours); 4=completely disabled, not capable of any self-care, totally confined to bed or chair. Higher scores signified =more functional impairment of a participant.
Time Frame: Baseline up to Cycle 43 (up to 1083 days)
Population: Safety analysis set included all enrolled participants who received at least 1 dose of axitinib or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
Participants
  0 | 39
  1 | 10
  2 | 0
  3 | 0
  4 | 0
  Missing | 3

9. Secondary Outcome: Objective Response Rate
Description: Objective response rate was defined as percentage of participants with confirmed complete response (CR) or confirmed partial response (PR), as assessed by response evaluation criteria in solid tumors (RECIST) version 1.1. Confirmed responses were those that persist on repeated imaging for at least 4 weeks after initial documentation of response. CR was defined as disappearance of all target lesions and the reduction in short axis of any pathological lymph nodes to <10 mm. PR was defined as a 30% or more decrease in the sum of longest dimensions of the target lesions, taking as reference the baseline sum of longest dimensions.
Time Frame: Baseline until disease progression or death due to any cause, up to a maximum of 1083 days
Population: Response evaluable analysis set included all participants who received study treatment with an adequate baseline tumor assessment (using standard RECIST version 1.1 criteria).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
percentage of participants | 73.1 [59.0 to 84.4]

10. Secondary Outcome: Duration of Response (DR)
Description: DR:date of first documentation of objective tumour response(OR) confirmed to date of first documentation of PD/death due to any cause,whichever occurred first.PD per RECIST 1.1:>=20%increase in sum of longest dimensions(LD) of target lesions,reference to smallest sum of LD recorded since treatment started/appearance of 1 or more new lesions/increase of at least 5mm addition to relative increase of 20%.DR calculated only for participants with confirmed OR.Participants lacking evaluation of tumour response after date of first study drug dose was censored on date of first dose unless death occurred prior to 18 weeks.If participants had at least 1 on-study assessment,PFS was censored on date of last evaluable tumour disease assessment documenting absence of PD for participants who were alive and progression free at time of analysis/had documentation of PD/death after>=2 consecutive missed tumour assessments/given anti-tumour treatment other than study drug prior to documented PD/death.
Time Frame: Baseline until disease progression or death due to any cause, up to a maximum of 1083 days
Population: Response evaluable analysis set included all participants who received study treatment with an adequate baseline tumor assessment (using standard RECIST version 1.1 criteria). Here, "N" signifies number of participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 38
months | 18.6 [15.1 to NA] — Number of participants with a confirmed objective response who subsequently progressed is too small to provide such summary statistics.

11. Secondary Outcome: Time to Response (TTR)
Description: TTR was defined as the time from first dose of study treatment to the first documentation of objective tumor response (CR or PR) that was subsequently confirmed.
Time Frame: Baseline until disease progression or death due to any cause, up to a maximum of 1083 days
Population: as for outcome 10
Measure: Median (Full Range); unit: months
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 38
months | 2.8 [0.7 to 15.2]

12. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS: time from date of first dose of study drug to the date of first documented PD or death on study due to any cause. PD as per RECIST v1.1 defined as at least a 20% increase in sum of longest dimensions of target lesions, reference to smallest sum of longest dimensions recorded since treatment started, or appearance of 1 or more new lesions or increase of at least 5 mm in addition to relative increase of 20%. Participants lacking an evaluation of tumor response after date of first study drug dose had event time censored on date of first dose unless death occurred prior to 18 weeks. If participants had at least 1 on-study assessment, PFS data was censored on date of last evaluable tumor disease assessment documenting absence of PD for participants who were alive and progression free at the time of analysis or had documentation of PD or had death after >=2 consecutive missed tumor assessments or were given anti-tumor treatment other than study drug prior to documented PD or death.
Time Frame: Baseline until disease progression or death due to any cause, up to a maximum of 1083 days
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
months | 20.9 [15.4 to NA] — Upper limit of 95% CI was not reached since a large proportion of participants in the analysis set had their PFS data censored and there were insufficient number of participants with events to calculate the full 95% CI.

13. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose of study drug to the date of death due to any cause. For participants still alive at the time of analysis, the OS time was censored on the last date the participants were known to be alive.
Time Frame: Baseline until disease progression or death due to any cause, up to a maximum of 1552 days
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
months | NA [43.7 to NA] — Median and upper limit for 95% CI could not be estimated because there were insufficient number of participants with event.

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Axitinib
Time Frame: Dose Finding Phase:Pre-dose,1,2,3,4,6,8 hours (hrs) post-dose on Day 7 of Lead-in (7 days prior Cycle 1 Day 1), Cycle 7 Day 1;Dose Expansion Phase:Pre dose,1,2,3,4,6,8 hrs post dose on Day 7 of Lead-in (7 days prior Cycle 1 Day 1), Cycle 7 Day 1
Population: Pharmacokinetic (PK) parameter analysis population included all treated participants who had at least 1 of the PK parameters of interest of any of the study drugs. Here "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure and "Number Analyzed" = participants evaluable for specific rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg: Participants with no prior systemic treatment for advance cancer, received axitinib 5 mg twice daily orally in combination with pembrolizumab (MK-3475) 2 mg/kg of body weight intravenous infusion every 3 weeks up to a maximum of 6 months in dose finding phase (each cycle of 21 days or lead-in day 21). Participants received axitinib up to a maximum of 64 cycles and pembrolizumab up to 56 cycles in dose expansion phase (each cycle of 21 days or lead-in day 21) until documented disease progression or unacceptable toxicity or study discontinuation criteria were met.
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 10
nanogram per milliliter (ng/mL)
  Dose finding phase: Day 7 of Lead-in | 46.58 (58)
  Dose finding phase: Day 1 of cycle 7: number analyzed (Participants) | 5
  Dose finding phase: Day 1 of cycle 7 | 36.57 (31)
  Dose expansion phase: Day 7 of Lead-in: number analyzed (Participants) | 9
  Dose expansion phase: Day 7 of Lead-in | 24.83 (85)
  Dose expansion phase: Day 1 of cycle 7: number analyzed (Participants) | 6
  Dose expansion phase: Day 1 of cycle 7 | 22.65 (51)

15. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Axitinib
Time Frame: Dose Finding Phase:Pre-dose, 1, 2, 3, 4, 6, 8 hrs post-dose on Day 7 of Lead-in (7 days prior Cycle 1 Day 1), Cycle 7 Day 1; Dose Expansion Phase:Pre-dose, 1, 2, 3, 4, 6, 8 hrs post-dose on Day 7 of Lead-in (7 days prior Cycle 1 Day 1), Cycle 7 Day 1
Population: PK parameter analysis population included all treated participants who had at least 1 of the PK parameters of interest of any of the study drugs. Here "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure and "Number Analyzed" = participants evaluable for specific rows.
Measure: Median (Full Range); unit: hour
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 10
hour
  Dose finding phase: Day 7 of Lead-in | 2.00 [1.00 to 4.00]
  Dose finding phase: Day 1 of cycle 7: number analyzed (Participants) | 5
  Dose finding phase: Day 1 of cycle 7 | 3.00 [3.00 to 4.00]
  Dose expansion phase: Day 7 of Lead-in: number analyzed (Participants) | 9
  Dose expansion phase: Day 7 of Lead-in | 2.00 [0.000 to 3.00]
  Dose expansion phase: Day 1 of cycle 7: number analyzed (Participants) | 6
  Dose expansion phase: Day 1 of cycle 7 | 2.00 [1.00 to 4.00]

16. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUC 0-12) of Axitinib
Time Frame: Dose Finding Phase:Pre-dose, 1, 2, 3, 4,6,8, 12 hrs post-dose on Day 7 of Lead-in (7 days prior Cycle 1 Day 1), Cycle 7 Day 1; Dose Expansion Phase:Pre-dose, 1,2,3,4,6,8,12 hrs post-dose on Day 7 of Lead-in (7 days prior Cycle 1 Day 1), Cycle 7 Day 1
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 10
nanogram*hour per milliliter (ng*hr/mL)
  Dose finding phase: Day 7 of Lead-in | 199.1 (46)
  Dose finding phase: Day 1 of cycle 7: number analyzed (Participants) | 5
  Dose finding phase: Day 1 of cycle 7 | 219.4 (12)
  Dose expansion phase: Day 7 of Lead-in: number analyzed (Participants) | 9
  Dose expansion phase: Day 7 of Lead-in | 92.99 (142)
  Dose expansion phase: Day 1 of cycle 7: number analyzed (Participants) | 6
  Dose expansion phase: Day 1 of cycle 7 | 116.9 (50)

17. Secondary Outcome: Apparent Oral Clearance (CL/F) of Axitinib
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes).
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 10
liter per hour (L/hr)
  Dose finding phase: Day 7 of Lead-in | 25.11 (46)
  Dose finding phase: Day 1 of cycle 7: number analyzed (Participants) | 5
  Dose finding phase: Day 1 of cycle 7 | 22.79 (12)
  Dose Expansion Phase: Day 7 of Lead-in: number analyzed (Participants) | 9
  Dose Expansion Phase: Day 7 of Lead-in | 53.77 (142)
  Dose expansion phase: Day 1 of cycle 7: number analyzed (Participants) | 6
  Dose expansion phase: Day 1 of cycle 7 | 42.79 (50)

18. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Axitinib
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 6
liter
  Dose finding phase: Day 7 of Lead-in | 85.12 (36)
  Dose finding phase: Day 1 of cycle 7: number analyzed (Participants) | 1
  Dose finding phase: Day 1 of cycle 7 | 50.91
  Dose Expansion Phase: Day 7 of Lead-in: number analyzed (Participants) | 5
  Dose Expansion Phase: Day 7 of Lead-in | 245.8 (50)
  Dose expansion phase: Day 1 of cycle 7: number analyzed (Participants) | 1
  Dose expansion phase: Day 1 of cycle 7 | 225.5

19. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) of Pembrolizumab (MK-3475)
Time Frame: Day 1 of Cycle 1 up to Day 21 of Cycle 56 (up to 1176 days)
Population: PK parameter analysis population included all treated participants who had at least 1 of the PK parameters of interest of any of the study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 52
Participants | 3

20. Secondary Outcome: Number of Participants With Programmed Death-Ligand 1 (PD-L1) Tumor Proportion Score
Description: PD-L1- tumor proportion score was defined as the percentage of viable tumor cells showing partial or complete membrane staining at any intensity. Participants with positive or negative scores were reported. PD-L1 negative: if tumor proportion score was less than 1%; PD-L1 positive: if the tumor proportion score greater than or equal to 1%.
Time Frame: Baseline up to Cycle 43 (up to 1083 days)
Population: Tumor biomarker analysis set included all treated participants who had at least one screening biomarker assessment, and had received at least one dose of any study drug. Here, "N" signifies number of participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 44
Participants
  Positive Score | 9
  Negative Score | 34
  Missing | 1

21. Secondary Outcome: Number of Participants With Vascular Endothelial Growth Factor A (VEGF-A) Tumor Proportion Score
Description: Vascular Endothelial Growth Factor (VEGF) promotes cancer progression by inducing angiogenesis via VEGF receptors, signals directly through receptors VEGFR-1 and VEGFR-2. Change in biomarkers related to VEGFR signal transduction pathways after axitinib treatment was assessed. Plasma VEGF concentration evaluations were performed using samples from peripheral blood plasma, bone marrow aspirate, bone marrow (Core) biopsy and bone marrow clot. The VEGFR, axitinib and mechanistic target of rapamycin inhibitor everolimus are used individually in subsequent lines of therapy for advanced clear cell renal cell carcinoma (ccRCC).
Time Frame: Baseline up to Cycle 64 (up to 1344 days)
Population: PDL1 analyses didn't find any statistically significant associations between PDL1 status and response, hence data for this outcome measure (a sub-analyses on PDL1 positive participants) was not further collected and analyzed.
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 0

22. Secondary Outcome: Concentration of Vascular Endothelial Growth Factor A (VEGF-A) in Serum
Description: Vascular endothelial growth factor (VEGF) promotes cancer progression by inducing angiogenesis via VEGF receptors, signals directly through receptors VEGFR-1 and VEGFR-2. Change in biomarkers related to VEGFR signal transduction pathways after axitinib treatment was assessed. Mononuclear (MNC) cell VEGF receptor expression and phosphorylation was assessed by in situ western blot analysis. VEGFR-1 and VEGFR-2 evaluations were performed using samples from peripheral blood plasma, bone marrow aspirate, bone marrow (Core) biopsy and bone marrow clot. The VEGFR, axitinib and mechanistic target of rapamycin inhibitor everolimus are used individually in subsequent lines of therapy for advanced clear cell renal cell carcinoma (ccRCC).
Time Frame: Baseline, Day 1 of Cycle 2 Pre-dose, Post end of treatment or Withdrawal whichever came first (maximum of 1344 days)
Population: Tumor biomarker analysis set included all treated participants who had at least one screening biomarker assessment, and had received at least one dose of any study drug. Here "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: picogram per millilitre (pg/mL)
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 51
picogram per millilitre (pg/mL)
  Baseline | 315.2 (286.6)
  Cycle 2 Day 1: number analyzed (Participants) | 49
  Cycle 2 Day 1 | 432.1 (315.0)
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 383.6 (360.4)

23. Secondary Outcome: Concentration of Vascular Endothelial Growth Factor Receptor 2 (VEGFR2) in Serum
Description: as for outcome 22
Time Frame: Baseline, Day 1 of Cycle 2 Pre-dose, Post end of treatment or Withdrawal whichever came first (maximum of 1344 days)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 51
nanogram per milliliter (ng/mL)
  Baseline | 4.11 (1.27)
  Cycle 2 Day 1: number analyzed (Participants) | 49
  Cycle 2 Day 1 | 3.07 (0.93)
  End of treatment: number analyzed (Participants) | 35
  End of treatment | 3.69 (1.41)

24. Secondary Outcome: Concentration of Interleukin 8 (IL-8) in Serum
Time Frame: Baseline, Day 1 of Cycle 2 Pre-dose, Post end of treatment or Withdrawal whichever came first (maximum of 1344 days)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
Number analyzed (Participants) | 51
mmol/L
  Baseline | NA (NA) — Data could not be estimated as concentration of IL-8 was less than lower limit of quantification.
  Cycle 2 Day 1: number analyzed (Participants) | 49
  Cycle 2 Day 1 | NA (NA) — Data could not be estimated as concentration of IL-8 was less than lower limit of quantification.
  End of treatment: number analyzed (Participants) | 35
  End of treatment | NA (NA) — Data could not be estimated as concentration of IL-8 was less than lower limit of quantification.

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (approximately up to 1552 days)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study. All treatment emergent AEs and non SAEs were collected and reported.
Arm/Group | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg
All-Cause Mortality (participants affected / at risk) | 14/52
Serious Adverse Events (participants affected / at risk) | 29/52
Other Adverse Events (participants affected / at risk) | 52/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg (N=52)
Atrial fibrillation (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Periorbital oedema (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Autoimmune colitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 6
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hepatotoxicity (Hepatobiliary disorders) | 1
Device related infection (Infections and infestations) | 1
Perineal abscess (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Embolism (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1
Pyelonephritis (Infections and infestations) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib 5 mg + Pembrolizumab (MK-3475) 2 mg (N=52)
Anaemia (Blood and lymphatic system disorders) | 11
Polycythaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Bradycardia (Cardiac disorders) | 4
Palpitations (Cardiac disorders) | 3
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Ear discomfort (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 3
Excessive cerumen production (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hyperthyroidism (Endocrine disorders) | 7
Hypothyroidism (Endocrine disorders) | 23
Thyroiditis (Endocrine disorders) | 1
Dry eye (Eye disorders) | 2
Erythema of eyelid (Eye disorders) | 2
Eye pain (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Periorbital oedema (Eye disorders) | 1
Vision blurred (Eye disorders) | 4
Visual impairment (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 14
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 4
Aerophagia (Gastrointestinal disorders) | 1
Buccal mucosal roughening (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 19
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 44
Dry mouth (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 10
Dysphagia (Gastrointestinal disorders) | 3
Faeces discoloured (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 6
Gastric ulcer (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5
Gingival disorder (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 5
Glossodynia (Gastrointestinal disorders) | 5
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 3
Hiatus hernia (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 23
Odynophagia (Gastrointestinal disorders) | 2
Oedema mouth (Gastrointestinal disorders) | 1
Oral discomfort (Gastrointestinal disorders) | 2
Oral disorder (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 13
Plicated tongue (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 8
Tongue discomfort (Gastrointestinal disorders) | 1
Tongue disorder (Gastrointestinal disorders) | 1
Tongue erythema (Gastrointestinal disorders) | 1
Tongue geographic (Gastrointestinal disorders) | 1
Tongue oedema (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 15
Asthenia (General disorders) | 2
Catheter site erythema (General disorders) | 1
Catheter site haematoma (General disorders) | 1
Catheter site oedema (General disorders) | 1
Chest pain (General disorders) | 2
Chest discomfort (General disorders) | 2
Chills (General disorders) | 7
Early satiety (General disorders) | 1
Face oedema (General disorders) | 1
Facial pain (General disorders) | 1
Fatigue (General disorders) | 42
Gait disturbance (General disorders) | 2
Hernia (General disorders) | 1
Influenza like illness (General disorders) | 5
Localised oedema (General disorders) | 2
Mucosal inflammation (General disorders) | 5
Non-cardiac chest pain (General disorders) | 2
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 11
Pain (General disorders) | 4
Peripheral swelling (General disorders) | 3
Pyrexia (General disorders) | 6
Cholecystitis acute (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Contrast media allergy (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 2
Abscess jaw (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Candida infection (Infections and infestations) | 3
Catheter site pustule (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Gingivitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Lip infection (Infections and infestations) | 2
Localised infection (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oropharyngitis fungal (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Parvovirus infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 2
Sinusitis bacterial (Infections and infestations) | 1
Skin candida (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 10
Urinary tract infection (Infections and infestations) | 4
Vulvovaginal mycotic infection (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 3
Ligament sprain (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Venous injury (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time abnormal (Investigations) | 1
Activated partial thromboplastin time prolonged (Investigations) | 5
Alanine aminotransferase increased (Investigations) | 21
Aspartate aminotransferase increased (Investigations) | 18
Bacterial test positive (Investigations) | 4
Blood alkaline phosphatase (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 6
Blood cholesterol increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 16
Blood phosphorus increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 2
Blood uric acid increased (Investigations) | 2
Cortisol decreased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 3
Haemoglobin increased (Investigations) | 3
International normalised ratio increased (Investigations) | 3
Liver function test increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 3
Neutrophil count increased (Investigations) | 1
Platelet count decreased (Investigations) | 8
Transaminases increased (Investigations) | 2
Weight decreased (Investigations) | 18
Weight increased (Investigations) | 4
White blood cell count decreased (Investigations) | 5
White blood cell count increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 23
Dehydration (Metabolism and nutrition disorders) | 7
Gout (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 7
Hypermagnesaemia (Metabolism and nutrition disorders) | 3
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 8
Hyponatraemia (Metabolism and nutrition disorders) | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 18
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Myositis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 2
Balance disorder (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 16
Dysgeusia (Nervous system disorders) | 11
Head discomfort (Nervous system disorders) | 1
Headache (Nervous system disorders) | 17
Hyperaesthesia (Nervous system disorders) | 1
Loss of proprioception (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 5
Neuralgia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 9
Presyncope (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 7
Confusional state (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 9
Libido decreased (Psychiatric disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 8
Micturition urgency (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 18
Cystocele (Reproductive system and breast disorders) | 1
Genital rash (Reproductive system and breast disorders) | 1
Penile pain (Reproductive system and breast disorders) | 1
Rectocele (Reproductive system and breast disorders) | 1
Uterine prolapse (Reproductive system and breast disorders) | 1
Vulval disorder (Reproductive system and breast disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 25
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14
Oropharyngeal cobble stone mucosa (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4
Blister (Skin and subcutaneous tissue disorders) | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 12
Erythema (Skin and subcutaneous tissue disorders) | 4
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 4
Nail ridging (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 19
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 12
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 14
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10
Rash papular (Skin and subcutaneous tissue disorders) | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Central venous catheterisation (Surgical and medical procedures) | 1
Embolism (Vascular disorders) | 1
Flushing (Vascular disorders) | 3
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 28
Hypotension (Vascular disorders) | 8
Labile blood pressure (Vascular disorders) | 1
Thrombophlebitis superficial (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Blepharitis (Eye disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Ill-defined disorder (General disorders) | 1
Prolapse (General disorders) | 1
Swelling (General disorders) | 1
Cystitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Tooth abscess (Infections and infestations) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 1
Activated partial thromboplastin time (Investigations) | 1
Bilirubin urine (Investigations) | 1
Blood creatine increased (Investigations) | 1
Blood phosphorus decreased (Investigations) | 1
Blood potassium decreased (Investigations) | 1
Blood uric acid abnormal (Investigations) | 1
Pancreatic enzymes decreased (Investigations) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Taste disorder (Nervous system disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Central venous catheter removal (Surgical and medical procedures) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT02133742/Prot_002.pdf
  • Statistical Analysis Plan (2015-07-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT02133742/SAP_001.pdf